CLINICAL TRIAL: NCT04093830
Title: Advantages of Bimodal Stimulation Compared to Unilateral Cochlear Implant Use in Children With Hearing Loss
Brief Title: Bimodal Stimulation Compared to Unilateral Cochlear Implant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Rizk Fam, Resident doctor -Assiut university hospital-Assiut, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: bimodal hearing
Record Dates: First submitted 2019-09-06; First posted 2019-09-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Hearing Impaired Children
Keywords: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pre-lingually deafened children with cochlear implant (Experimental): pre-lingually deafened children with cochlear implant who continuously used bimodal hearing.
  Interventions: Device: hearing aid

INTERVENTIONS:
Device: hearing aid — hearing aid can be used in their non- implanted ear with residual hearing

SUMMARY:
The majority of studies about bimodal hearing advantages have been conducted on adults but scant relevant studies into pediatric users, therefore more comparative studies are required to compare the effect of bimodal stimulation to unilateral cochlear implant use in children with severe to profound sensori-neural hearing loss .

DETAILED DESCRIPTION:
There are now many recipients of unilateral cochlear implants who have usable residual hearing in the non-implanted ear. To avoid auditory deprivation and to provide binaural hearing, a hearing aid or a second cochlear implant can be fitted to that ear. When bilateral cochlear implant cannot be used for patients with bilateral hearing impairment, a hearing aid can be used in their non- implanted ear with residual hearing. This is because patients with bilateral hearing loss need bilateral stimulation to develop the neural pathway required for central processing of binaural hearing.

ELIGIBILITY:
Inclusion Criteria:

1. The lack of middle-ear infection.
2. Normative intelligence.
3. The lack of auditory neuropathy disorder .
4. Residual hearing in the non-implanted ear.

Exclusion Criteria:

1. Middle ear infection..
2. Below average intelligence.
3. Auditory neuropathy disorder.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Comparison the audiometric thresholds in bimodal fitting users condition and cochlear implant alone condition | Baseline
  By using pure tone and speech audiometer the pure tone audiometry will be done in the free ﬁeld with a speaker at 0° azimuth and the mean threshold in speech frequencies of 0.5, 1, 2 and 4 kilohertz will be determined.
Comparison between speech discrimination score in bimodal fitting condition and cochlear implant alone condition. | Baseline
  The speech discrimination score is a measure as a percentage of words from a standardized list presented at suprathreshold levels that are recognized and repeated by the patient.
  a higher score on the speech discrimination test is better
  Interpreting speech discrimination score :
  100-90% Means Excellent or Normal speech discrimination score, 89-75% Means Good speech discrimination score, 74-60% Means Fair speech discrimination score, 59-50 % Means Poor speech discrimination score& <50% Means Very Poor speech discrimination score.
Evaluation of speech perception ability in noise under bimodal fitting a condition and cochlear implant alone condition | Baseline
  By speech perception in noise (SPIN) test using Compact disc on compact discs player.
Comparison of early speech perception in bimodal fitting condition and cochlear implant alone condition | Baseline
  The test will be done starting from a low level using the manual and standard scoring forms of Early speech perception test ( ESP) by using : Compact disc , full-color picture cards, Toys ,digitally remastered sounds, and an All Words menu
Comparison between the speech reception threshold in bimodal fitting condition and cochlear implant alone condition. | Baseline
  Speech reception threshold is the minimum intensity in decibels at which a patient can understand 50% of spoken words from a closed set list of disyllabic words

CONTACTS AND LOCATIONS:
Overall Officials: Enass S Mohamed, Professor, Principal Investigator — Professor of Audio-vestibular medicine,Assiut University,Egypt.

REFERENCES:
- [Background] Dorman MF, Gifford RH, Spahr AJ, McKarns SA. The benefits of combining acoustic and electric stimulation for the recognition of speech, voice and melodies. Audiol Neurootol. 2008;13(2):105-12. doi: 10.1159/000111782. Epub 2007 Nov 29. PMID 18057874
- [Background] Kokkinakis K, Pak N. Binaural advantages in users of bimodal and bilateral cochlear implant devices. J Acoust Soc Am. 2014 Jan;135(1):EL47-53. doi: 10.1121/1.4831955. PMID 24437856
- [Background] Tao DD, Liu JS, Yang ZD, Wilson BS, Zhou N. Bilaterally Combined Electric and Acoustic Hearing in Mandarin-Speaking Listeners: The Population With Poor Residual Hearing. Trends Hear. 2018 Jan-Dec;22:2331216518757892. doi: 10.1177/2331216518757892. PMID 29451107